CLINICAL TRIAL: NCT03713814
Title: Effects of an Exercise Protocol for Pilots With Back Pain.
Brief Title: Exercise Protocol for Pilots With Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor of Physiotherapy, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSLD2018
Record Dates: First submitted 2018-10-09; First posted 2018-10-22 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Low Back Pain
Keywords: Electromyography; Exercise therapy; Muscle Strength Dynamometer; Pilots; Back Pain
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 8-week exercise program, three times a week, during 45 minutes each section. Exercises for strength, endurance and mobility of the spine using pilates´ball and mat.
  Interventions: Other: Exercise
- Control group (No Intervention): After the 8 weeks of intervention, the pilots will receive explanation and handbook demonstration of the same exercises.

INTERVENTIONS:
Other: Exercise — 8-week exercise program, three times a week, during 45 minutes each section. Exercises for strength, endurance and mobility of the spine using pilates´ball and mat.
  The researcher will explain, demonstrate and supervise the participants. It will start with 10 minutes of warming-up using a ergometer bicycle, followed by the mat exercises. Some of these will require motor control with mobility, others will require isometry, or concentric and eccentric phases with progression of eccentric phase timing.
  Arms: Experimental Group

SUMMARY:
It is known that the low back pain can cause discomfort and deconcentration during the flight, requests for abstention of flight, fear in the aviators about the future in case of illness and economic damages to the country. However, there are few studies about the incidence, prevalence or risk factors associated with low back pain in Brazilian air force pilots. Also, the literature lacks further randomized controlled studies about interventions, leaving a huge field to be explored in future research.

Objectives: This study to analyze the chronic effects of an exercise protocol on lumbar pain in Brazilian Air Force pilots.

Materials and methods: The study is a blind and randomized clinical trial, in which a protocol of strength and lumbar resistance exercises will be tested. The volunteers will be: 20 fighter instructors with intermittent low back pain. Such volunteers will be recruited in a non-probabilistic manner for convenience. Moreover, they will be randomly distributed through www.randomization.com to form two groups with 10 members each: experimental group (EG), where they will participate in an exercise program three times a week for 8 weeks; and the control group (CG), in which they will receive explanation and handbook demonstration of the same exercises (Appendix 1) - after 8 weeks of intervention and after being reevaluated.

The study will be performed at the city of Natal/ Rio Grande do Norte. The evaluation will consist of an evaluation form with personal data, anthropometric data, occupational information, health history, physical exercise pattern and pain information, quantified by Visual Analog Pain Scale. In addition, the Oswestry questionnaire will be administered to assess lumbar function and the Nordic Questionnaire to assess musculoskeletal changes. Also, will be done: postural evaluation, using a postural evaluation software (SAPO); assessment of lumbar range of motion, using an IPHONE app called iHandy Level; Magnetic Resonance Imaging of the spine; dynamometry to measure the trunk extension force, flexion with rotation and lateral bridge, using the manual dynamometer Lafayette® - model 01165, USA; and resistance test of trunk stabilizing muscles. Magnetic resonance imaging will be done at the Onofre Lopes University Hospital. The project will be submitted to the Research Ethics Committee of the Federal University of Rio Grande do Norte through the national interface "Plataforma Brasil". The study will also be registered on the international clinical trial platform, ClinicalTrials.gov.

Data analysis: The Statistical Package for Social Science (SPSS) software will be used in the analysis. The normality of data distribution and the homogeneity of the variances will be verified by the Kolmogorov-Smirnov (K-S) and Levine tests, respectively. If there is a normal distribution, the descriptive statistics will be performed through means and standard deviations. Significance level adopted: 5% (P <0.05). The paired t test was used for the comparisons between the measurements obtained in the pre and post 2 month evaluations, and for the comparison between the groups (CG and EG), the unpaired t test. If the data do not present a normal distribution, the Friedman test will be used for comparisons of the measures of the evaluations in each group and the Kruskal-Wallis test for comparisons between the groups (CG and EG).

ELIGIBILITY:
Inclusion Criteria:

* Subject is fight pilot.
* Subject is flight instructor from the Brazilian Air Force.

Exclusion Criteria:

* Had not flown in the last 3 months
* History of acute lower back pain in the week of the evaluation
* Physical therapy during the study period
* History of heart disease or uncontrolled hypertension
* History of neurological disease
* History of rheumatic disease
* History of diabetes
* Do not perform the evaluation procedures correctly.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Change in number on Visual Analog Scale (VAS) of pain sensation in areas of the body (neck, shoulder, thoracic, low back spine, lower limbs) | Change from Baseline pain sensation at 8 weeks.
  Quantification in number on Visual Analog Scale (VAS) of pain sensation in areas of the body (neck, shoulder, thoracic, low back spine, lower limbs), considering the last week. In the VAS (minimum:0, maximum:10) zero means no pain, ten means the worse pain.
Change of disability of the Lower Back Muscles (LBM) at the day, measured by Oswestry Disability index (ODI) [Pain/Function of LBM] | Change from Baseline disability of the LBM at 8 weeks.
  Disability at the day measured by Oswestry Disability index (ODI). It has 10 six point scales. The sum of the 10 scores is expressed as a percentage of the maximum score. The first session gives the intensity of pain and the other 9 refer to the disabling effect on activities of daily living: personal care, weight lifting, sitting, walking, sleeping, sex life, social life, and traveling. The total score ranges from 0 (no disability) to 100 (disability maximum).

SECONDARY OUTCOMES:
BMI in kg/m^2 | Baseline.
  Weight and height will be combined to report BMI in kg/m^2.
Accumulated hours of flight | Baseline .
  Accumulated hours of flight (from the beginning of the career until today).
Presence of cervical and lumbar musculoskeletal injuries by using Magnetic Resonance Imaging assessment | Baseline.
  Presence of cervical and lumbar musculoskeletal injuries by using Magnetic Resonance Imaging assessment, evaluated by two physicians. The pilots will be directed to the Diagnostic Center by Image at the University Hospital Onofre Lopes (Natal-Rio Grande do Norte state,Brazil), where they will make the exams. The results will be referred by physicians to the researchers.
Change of the postural pattern | Change from Baseline Postural Evaluation at 8 weeks.
  Clinical evaluation of postural pattern by a physical therapist using the postural evaluation software (SAPO).
Assessment of lumbar spine range of motion. | Change from Baseline Strength of LBM at 8 weeks.
  The Iphone app called Ihandy level will be used by a physiotherapist in order to assess the range of motion of the lumbar spine in four movements: flexion, extension, right tilt and left tilt. The angles data will be recorded.
Change of Maximal Voluntary Isometric Contraction (MVIC) of Lower Back Muscles (LBM) measured in Newtons | Change from Baseline Strength of LBM at 8 weeks.
  Maximal Voluntary Isometric Contraction (MVIC) of Lower Back Muscles (LBM) to be assessed similar to the protocol assessed by Nakagawa et al., 2015.
  The individual wil be requested to sustain isometry during 5 seconds, of 3 different positions of the trunk: flexion with rotation for the external oblique muscle MVIC measure and extension of trunk for iliocostalis MVIC measure. The testing order was randomised to account for ordering bias. It will be used the handheld dynamometer - Lafayette for the measure and it will be recorded in Newtons. The greatest measure will be chosen.
Change in number of affirmative answers for presence of referred musculoskeletal disorders, measured by Nordic Musculoskeletal Questionnaire. | Change from Baseline Presence of musculoskeletal disorders at 8 weeks.
  Nordic Musculoskeletal Questionnaire - the aim of the questionnaire is to evaluate musculoskeletal problems in an ergonomic approach. The first part of the instrument consists of questions related to parts of the human body that correspond to nine anatomical areas (3 upper limbs, 3 lower limbs, 3 - trunk), marked in an illustration of the human body seen from the back. The questions are organized as follows: weekly and annual prevalence; functional disability; and health care research in the last 12 months. The instrument will be answered by the pilot individually; scribbling yes or no to each question
Change of time in seconds of sustained isometry in 3 positions of trunk (flexion, extension and side-bridge) [Endurance of Lower Back Muscles (LBM)] | Change from Baseline Endurance of LBM at 8 weeks.
  Endurance of LBM will be measured by the seconds of sustained isometry in 3 position (flexion with rotation, extension and side-bridge). The time will be counted by clock chronometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

REFERENCES:
- [Derived] Mendes PRF, Gomes SRA, Costa LDO, Liguori ADAL, Bulhoes LCC, Brasileiro JS. Core stabilisation exercises reduce chronic low back pain in Air Force fighter pilots: a randomised controlled trial. BMJ Mil Health. 2024 Jan 25;170(1):31-36. doi: 10.1136/bmjmilitary-2021-002005. PMID 35470256